CLINICAL TRIAL: NCT00768196
Title: Prevalence of EED and Quality of Life Evaluated by Gastroesophageal Reflux Disease (GERD)-Q in Korean GERD Patients
Acronym: Preedom
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Other Study IDs: NIS-GKR-DUM-2008/1
Record Dates: First submitted 2008-10-01; First posted 2008-10-07 (Estimated); Last update posted 2010-12-07 (Estimated); Status verified 2010-12

CONDITIONS: Gastroesophageal Reflux Disease
Keywords: GERD; Korea; typical symptom; quality of life; Naturalistic; epidemiological
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to asses the EED symptom prevalence in Koran GERD patients with typical reflux symptom and to evaluate quality of life with the scales including Gerd Q.

ELIGIBILITY:
Inclusion Criteria:

* GERD patients who have experienced heartburn or acid regurgitation during past 7 days
* GERD patients who have already undergone endoscopy before enrolment

Exclusion Criteria:

* Involvement in the planning and conduct of the programme
* The person who took the medicine such as PPI or H2RA during the last 7 days
* Severe systemic disease

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: general hospital sample
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2008-09; Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
The primary variable is the total rate of GERD patients who had EED symptom and effect on their quality of life.

SECONDARY OUTCOMES:
The secondary variable is the comparison of the EED symptom frequency in ERD and NERD patients.

CONTACTS AND LOCATIONS:
Overall Officials: Joon-Woo Bahn, Study Director — AstraZeneca Korea
Locations (4):
- South Korea (4):
  - Research Site, Cheonan, Chungcheongnam-do
  - Research Site, Seoul, Kyungkido
  - Research Site, Sungnam, Kyungkido
  - Research Site, Suwon, Kyungkido